CLINICAL TRIAL: NCT03641014
Title: Sequential pH Effect on Blastocyst Formation Rate
Brief Title: Whether Using Sequential pH Would Improve Human Blastocyst Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other); Quena IVF Centre (Unknown)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-Sequential pH
Record Dates: First submitted 2018-08-10; First posted 2018-08-21 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential pH culture (7.23 then 7.35) (Experimental): A split embryo at day 3 to continue culture at a pHe of 7.23±0.02 or to be cultured at a pH of 7.35±0.02 and monitor the effect on blastocyst development.
  Interventions: Other: pH Effect on blastocyst formation
- Continuously pH culture at 7.23 (No Intervention): Embryo culture from day 0 to 5 or 6 at 7.23

INTERVENTIONS:
Other: pH Effect on blastocyst formation — to investigate which pH is suitable for each stage of embryo development
  Arms: Sequential pH culture (7.23 then 7.35)

SUMMARY:
Any drift in extracellular pH (pHe) from the intercellular pH (pHi) could alter the mechanism regulating transporters and exchangers through the plasma membrane. This could lead to difficulty in restoring the physiological level of pHi. The critical stages that lack robust mechanism of regulating the pHi are the denuded oocyte, early stage of fertilization or a thawed embryo. This, in turn, could lead to a significant effect of the perturbations on embryo development. Convincing evidence regarding the optimal pHe for culturing human embryo is, so far, scanty and mostly anecdotal. The embryo has been reported to have a compensatory mechanism to grow at pHe between 7.0-7.4. Others have recommended that embryo need a sequential pH to viably grow suggesting that the post-genomic activation stage needs a slightly alkaline range of pH. However, whether this holds true remains to be examined.

ELIGIBILITY:
Inclusion Criteria:

* ICSI cycles

Exclusion Criteria:

* No exclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1312 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Ongoing Pregnancy rate | 12 weeks
  women with continued pregnancy at week 12 of gestation

SECONDARY OUTCOMES:
rate of usable blastocysts | 6 days of culture
  number of blastocysts suitable for transfer on day 5 or 6
Blastocyst formation rate | 6 days of culture
  number of formed blastocyst per Fertilized oocyte
Clinical pregnancy rate | 3 months
  number of women with ultrasound detection of sacs with heartbeat per stimulated cycle
Implantation rate | 7 weeks
  number of sacs with a heartbeat

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Quena IVF Centre, Quena, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag

IPD SHARING:
Plan to Share IPD: No